CLINICAL TRIAL: NCT03250676
Title: A Phase 1-2 Multicenter, Open Label Trial of H3B-6545, a Covalent Antagonist of Estrogen Receptor Alpha, in Women With Locally Advanced or Metastatic Estrogen Receptor-positive, HER2 Negative Breast Cancer
Brief Title: Trial of H3B-6545, in Women With Locally Advanced or Metastatic Estrogen Receptor-positive, HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H3B-6545-A001-101; 2018-000570-29 (EudraCT Number)
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-03

CONDITIONS: Breast Neoplasms; Breast Cancer; Estrogen-receptor Positive Breast Cancer; Cancer, Breast; Breast Cancer Female; Breast Adenocarcinoma; Estrogen Receptor Positive Tumor; ER Positive
Keywords: estrogen receptor; H3B-6545; breast cancer; Endocrine Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — H3B-6545

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- H3B-6545 Arm 1: Dose escalation (Experimental)
  Interventions: Drug: H3B-6545
- H3B-6545 Arm 2: Phase 2 (Experimental)
  Interventions: Drug: H3B-6545

INTERVENTIONS:
Drug: H3B-6545 — Oral capsules by mouth once daily

SUMMARY:
The primary purpose of phase 1 portion of this study is to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of H3B-6545 in women with locally advanced or metastatic estrogen receptor (ER)-positive, human epidermal growth factor 2 (HER2)-negative breast cancer.

The primary purpose of phase 2 portion of this study is to estimate the efficacy of H3B-6545 in terms of best overall response rate, duration of response (DoR), clinical benefit rate (CBR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS) in all participants with ER-positive, HER2-negative breast cancer and in those with and without ER alpha mutation (including a clonal estrogen receptor 1 gene [ESR1] Y537S mutation).

ELIGIBILITY:
Inclusion Criteria:

1. Pre- or post-menopausal women.
2. ER-positive, HER2-negative breast cancer that is advanced or metastatic.
3. Progressed on prior therapy. Multiple prior lines of therapy allowed in Phase 1 and 2. Participants under amendment 6 (or subsequent amendments) must have received prior cyclin-dependent kinase (CDK4/6) inhibitor therapy. Up to one prior chemotherapy in the metastatic setting is allowed.
4. A recent archival tumor tissue obtained within 6 months prior to enrollment or a fresh tumor biopsy must be provided. A second biopsy after initiating trial therapy is not required.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
6. Adequate bone marrow and organ function.
7. Participants under amendment 6 (or subsequent amendments) must have measurable disease at baseline as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.
8. Participants under amendment 6 (or subsequent amendments) must have ESR1 Y537S mutation in absence of ESR1 D538G mutation as per the results of a central laboratory from a Nucleic Acids Whole Blood sample.

Exclusion Criteria:

1. Participants must have at least one measurable lesion.
2. Participant with inflammatory breast cancer.
3. Participant has received more than one prior chemotherapy regimen for metastatic disease (Phase 2 only).
4. Females of childbearing potential who are unable or unwilling to follow adequate contraceptive measures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (23):
  - Western Regional Medical Center, Inc., DBA Cancer Treatment Centers of America, Phoenix, Goodyear, Arizona
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado - Cancer Center, Aurora, Colorado
  - Holy Cross Hospital Inc, Fort Lauderdale, Florida
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Florida Cancer Specialists and Research Institute, Sarasota, Florida
  - Florida Cancer Specialists North, St. Petersburg, Florida
  - Southeastern Regional Medical Center, Inc., DBA Cancer Treatment Centers of America, Atlanta, Newnan, Georgia
  - Carle Cancer Center, Urbana, Illinois
  - Midwestern Regional Medical Center, Inc., DBA Cancer Treatment Centers of Americal, Chicago, Zion, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - University of North Carolina, Chapel Hill, North Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Parkland Health and Hospital System, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Tyler Oncology/Oncology PA, Tyler, Texas
  - Huntsman Cancer Institute at The University of Utah, Salt Lake City, Utah
- France (10):
  - Edog - Ico - Ppds, Angers
  - Hopital Jean Minjoz, Besançon
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Hôpital Saint Louis, Paris
  - Hôpital de la Pitié Salpétrière, Paris
  - EDOG - Centre Eugene Marquis Centre Regional de Lutte Contre Le Cancer - PPDS, Rennes
  - EDOG Institut de Cancerologie de l'Ouest - PPDS, Saint-Herblain
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - Institut Gustave Roussy, Villejuif
- United Kingdom (6):
  - The Royal Marsden NHS Foundation Trust, Chelsea, London
  - Velindre Cancer Centre, Cardiff
  - Barts Health NHS Trust, London
  - Sarah Cannon Research Institute, London
  - Christie Hospital, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

REFERENCES:
- [Derived] Furman C, Puyang X, Zhang Z, Wu ZJ, Banka D, Aithal KB, Albacker LA, Hao MH, Irwin S, Kim A, Montesion M, Moriarty AD, Murugesan K, Nguyen TV, Rimkunas V, Sahmoud T, Wick MJ, Yao S, Zhang X, Zeng H, Vaillancourt FH, Bolduc DM, Larsen N, Zheng GZ, Prajapati S, Zhu P, Korpal M. Covalent ERalpha Antagonist H3B-6545 Demonstrates Encouraging Preclinical Activity in Therapy-Resistant Breast Cancer. Mol Cancer Ther. 2022 Jun 1;21(6):890-902. doi: 10.1158/1535-7163.MCT-21-0378. PMID 35642432

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 39 investigative sites in the United States, France, and the United Kingdom from 23 Aug 2017 to 26 Oct 2023. This study was conducted in two parts: dose escalation and dose expansion.
Pre-assignment Details: In the dose escalation part, a total of 47 participants were enrolled and received the study treatment and 104 participants were enrolled in the dose expansion part and received the study treatment. A food-effect sub-study was conducted during the dose expansion phase, where a total of 18 participants (9 participants in each intervention sequence) received H3B-6545 under fed and fasted conditions in a cross-over manner and aided in evaluation of pharmacokinetic (PK) data.
Groups:
- Phase 1: Dose Escalation: H3B-6545 100 mg: Participants received H3B-6545 100 milligram (mg) capsule, orally, once daily (QD) in each 28-days cycle until disease progression, unacceptable toxicity, withdrawal of consent or study discontinuation.
- Phase 1: Dose Escalation: H3B-6545 200 mg: Participants received H3B-6545 200 mg capsule, orally, QD in each 28-days treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent or study discontinuation.
- Phase 1: Dose Escalation: H3B-6545 300 mg: Participants received H3B-6545 300 mg capsule, orally, QD in each 28-days treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent or study discontinuation.
- Phase 1: Dose Escalation: H3B-6545 450 mg; Phase 2: Dose Expansion: H3B-6545 450 mg: Participants received H3B-6545 450 mg capsule, orally, QD in each 28-days treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent or study discontinuation.
- Phase 1: Dose Escalation: H3B-6545 600 mg: Participants received H3B-6545 600 mg capsule, orally, QD in each 28-days treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent or study discontinuation.
Period: Overall Study
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1: Dose Escalation: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg | Phase 2: Dose Expansion: H3B-6545 450 mg
Started | 6 | 12 | 11 | 11 | 7 | 104
Food-effect Cohort - Fasted Then Fed (Food-effect Analysis Set (Phase 2): All participants who were assigned to the food-effect cohort and had sufficient PK data to derive at least 1 PK parameter.) | 0 | 0 | 0 | 0 | 0 | 9
Food-effect Cohort - Fed Then Fasted | 0 | 0 | 0 | 0 | 0 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 12 | 11 | 11 | 7 | 104
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 9
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0 | 3
Not completed — Withdrawal of consent | 0 | 0 | 2 | 0 | 0 | 2
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 4 | 12 | 9 | 7 | 4 | 88

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least one dose of study drug.
Groups:
- Phase 1: Dose Escalation: H3B-6545 100 mg: Participants received H3B-6545 100 mg capsule, orally, QD in each 28-days treatment cycle until disease progression, unacceptable toxicity, withdrawal of consent or study discontinuation.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1: Dose Escalation: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg | Phase 2: Dose Expansion: H3B-6545 450 mg | Total
Number analyzed (Participants) | 6 | 12 | 11 | 11 | 7 | 104 | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 7 | 8 | 3 | 61 | 90
  >=65 years | 3 | 4 | 4 | 3 | 4 | 43 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 12 | 11 | 11 | 7 | 104 | 151
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 0 | 5 | 7
  Not Hispanic or Latino | 6 | 10 | 11 | 11 | 7 | 98 | 143
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 5 | 7
  White | 6 | 9 | 10 | 11 | 7 | 84 | 127
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 0 | 12 | 14

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose-limiting Toxicities (DLTs)
Description: DLT was graded as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. DLTs were defined as the following events that occurred in Cycle 1, for which a causal relationship with the study drug could not be ruled out: febrile neutropenia; Grade 4 neutropenia that was not resolved within 7 days; Grade 4 thrombocytopenia; Grade 3 thrombocytopenia lasting greater than (>) 7 days or associated with clinically significant bleeding; Grade 4 vomiting and diarrhea; Grade 3 vomiting and diarrhea lasting >72 hours despite treatment; Grade 4 electrolyte abnormality or Grade 3 abnormality lasting >24 hours; Grade 3 or 4 serum creatinine or bilirubin increase; Grade 4 biochemistry or Grade 3 lasting >7 days; Grade 4 or Grade 3 or intolerable Grade 2 toxicities of any non-hematologic adverse event.
Time Frame: Cycle 1 (Cycle length=28 days)
Population: Dose evaluable set included all participants who were evaluated for DLTs in dose escalation part.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1: Dose Escalation: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 10 | 11 | 10 | 5
Participants | 0 | 0 | 0 | 0 | 2

2. Primary Outcome: Phase 1 and Phase 2: Objective Response Rate (ORR)
Description: ORR was assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as defined by the Investigator based on radiologic criteria. ORR was defined as the percentage of participants who achieved a best overall response of confirmed partial response (PR) or complete response (CR). CR was defined as disappearance of all target lesions, any pathological lymph nodes (whether target or non-target) with reduction in short axis to less than (<)10 millimeter (mm). PR was defined as at least a 30 percentage (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. As per planned analysis, pooled data for phase 1 and phase 2 for 450 mg dose was presented as enrolled participants in both the phases had similar demographics and disease characteristics.
Time Frame: Phase 1 and Phase 2: From the first dose of study drug to the first date of documentation of progressive disease (PD) or death, whichever occurred first (up to 33 months)
Population: Response-evaluable set included those participants who received at least 1 dose of study drug and had measurable disease at baseline and at least 1 post-baseline evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Phase 1 and Phase 2: H3B-6545 450 mg: In Phase 1 (dose-escalation) and Phase 2 (dose expansion), participants received H3B-6545 450 mg capsule, orally, QD in each 28-days treatment cycle until disease progression, unacceptable toxicity, or withdrawal of consent.
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 11 | 10 | 94 | 5
percentage of participants | 16.7 [0.4 to 64.1] | 9.1 [0.2 to 41.3] | 0 [0.0 to 30.8] | 20.2 [12.6 to 29.8] | 0 [0.0 to 52.2]

3. Primary Outcome: Phase 1 and Phase 2: Duration of Response (DoR)
Description: The DoR was assessed according to RECIST version 1.1. DoR was defined as the time from the date of the first documented CR/PR until the first documentation of disease progression or death, whichever comes first. CR was defined as disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. As per planned analysis, pooled data for phase 1 and phase 2 for 450 mg arm was presented as enrolled participants in both the phases had similar demographics and disease characteristics.
Time Frame: Phase 1 and Phase 2: From the first dose of study drug to the first date of documentation of PD or death, whichever occurred first (up to 33 months)
Population: Response-evaluable set included those participants who received at least 1 dose of study drug and had measurable disease at baseline and at least 1 post-baseline evaluation. Here, "Overall number of participants analyzed" signifies participants who had CR or/and PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 1 | 1 | 0 | 19 | 0
months | 7.95 [NA to NA] — Upper and lower range of 95% confidence interval (CI) could not be estimated due to insufficient events. | 6.05 [NA to NA] — Upper and lower range of 95% CI could not be estimated due to insufficient events. |  | 9.23 [5.88 to 20.24] |

4. Primary Outcome: Phase 1 and Phase 2: Disease Control Rate (DCR)
Description: The DCR was assessed according to RECIST version 1.1. DCR was defined as the percentage of participants who achieved best response of CR, PR, or stable disease (SD). CR was defined as disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (at least a 20% increase in the sum of diameters of target lesions) taking as reference the smallest sum diameters while on study. As per planned analysis, pooled data for phase 1 and phase 2 for 450 mg arm was presented as enrolled participants in both the phases had similar demographics and disease characteristics.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 11 | 10 | 94 | 5
percentage of participants | 100.0 [54.1 to 100.0] | 54.5 [23.4 to 83.3] | 30.0 [6.7 to 65.2] | 61.7 [51.1 to 71.5] | 40.0 [5.3 to 85.3]

5. Primary Outcome: Phase 1 and Phase 2: Clinical Benefit Rate (CBR)
Description: The CBR was assessed according to RECIST version 1.1. CBR defined as the percentage of participants with best overall response (BOR) of PR, CR, or durable SD (duration >=23 weeks). It was calculated for participants whose BOR was SD. CR defined as disappearance of all target lesions; any pathological lymph nodes (whether target or non-target) with reduction in short axis to <10 mm. PR defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (at least a 20% increase in the sum of diameters of target lesions) taking as reference the smallest sum diameters on study. As per planned analysis, pooled data for phase 1 and phase 2 for 450 mg arm was presented as enrolled participants in both the phases had similar demographics and disease characteristics.
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 11 | 10 | 94 | 5
percentage of participants | 83.3 [35.9 to 99.6] | 27.3 [6.0 to 61.0] | 20.0 [2.5 to 55.6] | 41.5 [31.4 to 52.1] | 40.0 [5.3 to 85.3]

6. Primary Outcome: Phase 1 and Phase 2: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose date to the date of the first documentation of PD or death whichever occurred first. PD defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum diameters while on study. As per planned analysis, pooled data for phase 1 and phase 2 for 450 mg arm was presented as enrolled participants in both the phases had similar demographics and disease characteristics.
Time Frame: as for outcome 3
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 12 | 11 | 115 | 7
months | 9.28 [7.43 to NA] — Upper range of 95% CI could not be estimated due to higher number (>50%) of censored participants. | 3.38 [1.31 to 7.75] | 1.84 [1.61 to 5.36] | 4.60 [3.52 to 6.67] | 2.76 [0.49 to 5.32]

7. Primary Outcome: Phase 1 and Phase 2: Overall Survival (OS)
Description: OS was defined as the time from first dose date to the date of death (event) or date last known alive (censored). As per planned analysis, pooled data for phase 1 and phase 2 for 450 mg arm was presented as enrolled participants in both the phases had similar demographics and disease characteristics.
Time Frame: Phase 1 and Phase 2: From the first dose of study drug to date of death or last known alive (up to 63 months)
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 12 | 11 | 115 | 7
months | 12.37 [7.43 to NA] — Upper range of 95% CI could not be estimated due to higher number (>50%) of censored participants. | 11.25 [1.87 to 40.41] | 13.50 [2.37 to 27.60] | 21.52 [16.56 to 25.46] | 5.32 [2.33 to 11.56]

8. Secondary Outcome: Phase 1 and 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: TEAE was defined per NCI CTCAE version 4.03 as an adverse event (AE) with an onset that occurred after receiving study drug. An AE was defined as any untoward medical occurrence in a participant administered an investigational product. An AE does not necessarily have a causal relationship with medicinal product. A serious adverse event (SAE) was defined as any AE if it resulted in death or life-threatening AE or required inpatient hospitalization or prolongation of existing hospitalization or resulted in persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions or was a congenital anomaly/birth defect. Pooled data from phase 1 and phase 2 was presented for 450 mg arm as enrolled participants in both the phases had similar demographics and disease characteristics with no major changes in inclusion/exclusion criteria as defined in the protocol.
Time Frame: From start of the study up to 74 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 12 | 11 | 115 | 7
Participants
  TEAEs | 6 | 12 | 11 | 115 | 7
  SAEs | 2 | 1 | 2 | 30 | 1

9. Secondary Outcome: Phase 1: (AUC0-t): Area Under the Plasma Concentration-time Curve From Time 0 Through the Last Measurable Point of H3B-6545
Description: AUC(0-t) was defined as the area under the plasma concentration-time curve from 0 time to last measurable point for H3B-6545.
Time Frame: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length = 28 days)
Population: PK analysis set included all participants who had received at least 1 dose of study drug H3B-6545 and had sufficient PK data to derive at least 1 PK parameter. Here, "number analyzed" signifies participants who were evaluable for specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/mL)
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1: Dose Escalation: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 12 | 11 | 11 | 7
hour*nanogram per milliliter (h*ng/mL)
  Cycle 1 Day 1 | 1680 (85.4) | 3310 (66.5) | 8520 (49.0) | 16200 (43.2) | 12600 (512)
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 10 | 11 | 10 | 2
  Cycle 1 Day 15 | 2590 (57.4) | 5200 (70.6) | 10700 (50.3) | 14100 (53.2) | 14900 (99.5)

10. Secondary Outcome: Phase 1: Cmax: Maximum Observed Plasma Concentration for H3B-6545
Description: Cmax was defined as the maximum plasma concentration for H3B-6545.
Time Frame: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length = 28 days)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1: Dose Escalation: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 12 | 11 | 11 | 7
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 178 (85.3) | 391 (55.7) | 879 (62.5) | 1500 (53.1) | 1490 (167)
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 10 | 11 | 10 | 2
  Cycle 1 Day 15 | 287 (31.3) | 605 (56.0) | 1200 (38.2) | 1410 (53.5) | 1310 (129)

11. Secondary Outcome: Phase 1: Tmax: Time of Maximum Observed Plasma Concentration of H3B-6545
Description: Tmax was defined as the time to reach maximum observed plasma concentration for H3B-6545.
Time Frame: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length = 28 days)
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1: Dose Escalation: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 12 | 11 | 11 | 7
hours
  Cycle 1 Day 1 | 3.05 [2.00 to 6.00] | 3.00 [2.00 to 6.17] | 3.97 [2.00 to 6.00] | 4.00 [2.00 to 10.00] | 4.00 [2.00 to 6.00]
  Cycle 1 Day 15: number analyzed (Participants) | 6 | 10 | 11 | 10 | 2
  Cycle 1 Day 15 | 2.00 [2.00 to 8.03] | 2.17 [2.00 to 6.00] | 4.00 [2.00 to 5.95] | 4.00 [1.00 to 8.00] | 5.00 [4.00 to 6.00]

12. Secondary Outcome: Phase 1: Rac (Cmax): Accumulation Ratio of Cmax for H3B-6545
Description: Accumulation ratio of Cmax was calculated as Cmax at Cycle 1 Day 15/Cmax at Cycle 1 Day 1.
Time Frame: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length = 28 days)
Population: PK analysis set included all participants who had received at least 1 dose of study drug H3B-6545 and had sufficient PK data to derive at least 1 PK parameter. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1: Dose Escalation: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 10 | 11 | 10 | 2
ratio | 1.61 (69.3) | 1.52 (80.6) | 1.37 (35.8) | 1.05 (42.1) | 0.598 (98.0)

13. Secondary Outcome: Phase 1: Rac (AUC0-24h): Accumulation Ratio of Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Postdose (AUC0-24h) for H3B-6545
Description: Rac (AUC0-24h) was calculated as AUC(0-24h) at Cycle 1 Day 15/AUC(0-24h) at Cycle 1 Day 1.
Time Frame: Cycle 1 Days 1 and 15: predose and up to 24 hours postdose (Cycle length = 28 days)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1: Dose Escalation: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 6 | 8 | 9 | 10 | 2
ratio | 1.52 (58.3) | 1.55 (77.8) | 1.23 (26.1) | 0.917 (48.5) | 0.646 (37.5)

14. Secondary Outcome: Phase 2: Relative Bioavailability (Food Effect) of H3B-6545 Assessed Using AUC(0-24h)
Description: Relative bioavailability based on food effect was calculated by taking ratio of AUC(0-24h) under fed condition divided by AUC(0-24h) under fasting condition. Data for the fasted and fed cohorts was collected on both Day 15 and Day 22 and was averaged.
Time Frame: Cycle 1 Days 15 and 22: predose and up to 24 hours postdose (Cycle length = 28 days)
Population: Food-effect analysis set included all participants who were assigned to the food-effect cohort and had sufficient PK data to derive at least 1 PK parameter. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Phase 2: Dose Expansion: H3B-6545 450 mg
Number analyzed (Participants) | 13
ratio | 1.53 [1.19 to 1.98]

15. Secondary Outcome: Phase 2: Relative Bioavailability (Food Effect) of H3B-6545 Assessed Using Cmax
Description: Relative bioavailability based on food effect was calculated by taking ratio of Cmax under fed condition divided by Cmax under fasting condition. Data for the fasted and fed cohorts was collected on both Day 15 and Day 22 and was averaged.
Time Frame: Cycle 1 Days 15 and 22: predose and up to 24 hours postdose (Cycle length = 28 days)
Population: Food-effect analysis set included all participants who were assigned to the food-effect cohort and had sufficient PK data to derive at least 1 PK parameter.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: ratio
Arm/Group | Phase 2: Dose Expansion: H3B-6545 450 mg
Number analyzed (Participants) | 18
ratio | 1.51 [1.20 to 1.90]

16. Secondary Outcome: Phase 2: Mean Change From Baseline in Endometrial Thickness Due to H3B-6545
Description: Participants with an intact uterus underwent transvaginal ultrasound to examine the effect of H3B-6545 on endometrial thickness. Baseline was defined as the last non-missing value before the first dose of study drug (Day 1). Mean change from baseline was calculated as post-baseline visit value minus baseline value.
Time Frame: Baseline, Week 12, Week 36 and Week 60
Population: Endometrium safety evaluable set included all participants with intact uteri at baseline, who received at least 1 dose of study drug and had ultrasound assessments at screening/baseline and three months after starting trial therapy. Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure and "Number analyzed" signifies participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Phase 2: Dose Expansion: H3B-6545 450 mg
Number analyzed (Participants) | 24
millimeter
  At Week 12: number analyzed (Participants) | 20
  At Week 12 | 4.079 (4.9659)
  At Week 36: number analyzed (Participants) | 7
  At Week 36 | 5.400 (6.9931)
  At Week 60: number analyzed (Participants) | 2
  At Week 60 | -0.050 (0.0707)

17. Secondary Outcome: Phase 2: Mean Change From Baseline in Uterine Volume Due to H3B-6545
Description: Participants with an intact uterus underwent transvaginal ultrasound to examine the effect of H3B-6545 on uterine volume. Baseline was defined as the last non-missing value before the first dose of study drug (Day 1). Mean change from baseline was calculated as post-baseline visit value minus baseline value.
Time Frame: Baseline, Week 12 and Week 36
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Phase 2: Dose Expansion: H3B-6545 450 mg
Number analyzed (Participants) | 24
milliliter
  At Week 12: number analyzed (Participants) | 21
  At Week 12 | 66.822 (63.7151)
  At Week 36: number analyzed (Participants) | 7
  At Week 36 | 41.083 (60.6320)

18. Secondary Outcome: Phase 1 and 2: Change From Baseline in Bone Turn-over Marker - Bone-specific Alkaline Phosphatase
Description: Blood samples were collected at indicated timepoint for evaluation of bone turn-over marker BSAP. Baseline is defined as the last non-missing value before the first dose of study drug (Day1). Change from baseline was calculated as post-baseline visit value minus baseline value. Pooled data from phase 1 and phase 2 was presented for 450 mg arm as enrolled participants in both the phases had similar demographics and disease characteristics with no major changes in inclusion/exclusion criteria as defined in the protocol.
Time Frame: Baseline (predose), Cycle 2 Day 15, Cycle 4 Day 1, and off-Treatment (up to 33 months) (Cycle length = 28 days)
Population: Bone turnover markers-evaluable set included participants who had baseline/screening assessments of bone turnover markers and at least 1 additional assessment at 6 and/or 12 weeks after starting trial therapy. Here, "number of participants analyzed" signifies participants who were evaluable for this outcome measure and "n" signifies participants who were evaluable for specified timepoints.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 0 | 3 | 3 | 75 | 3
units per liter (U/L)
  Cycle 2 Day 15 |  | -5.543 (14.7690) | 2.327 (4.5368) | 5.912 (40.7469) | -5.683 (5.4399)
  Cycle 4 Day 1: number analyzed (Participants) | 0 | 1 | 0 | 50 | 1
  Cycle 4 Day 1 |  | -0.390 (NA) — Standard deviation could not be estimated due to insufficient number of participants. |  | 0.381 (33.6782) | -0.900 (NA) — Standard deviation could not be estimated due to insufficient number of participants.
  Off-Treatment: number analyzed (Participants) | 0 | 0 | 0 | 23 | 0
  Off-Treatment |  |  |  | -4.469 (37.2991) |

19. Secondary Outcome: Phase 1 and 2: Change From Baseline in Bone Turn-over Marker - Amino-Terminal Propeptide of Type 1 Collagen (PINP)
Description: Blood samples were collected at indicated timepoint for evaluation of Bone turn-over marker PINP. Baseline is defined as the last non-missing value before the first dose of study drug (Day 1). Change from baseline was calculated as post-baseline visit value minus baseline value. Pooled data from phase 1 and phase 2 was presented for 450 mg arm as enrolled participants in both the phases had similar demographics and disease characteristics with no major changes in inclusion/exclusion criteria as defined in the protocol.
Time Frame: Baseline (predose), Cycle 2 Day 15, Cycle 4 Day 1, and off-Treatment (up to 33 months) (Cycle length = 28 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: micrograms per liter (mcg/L)
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 4 | 9 | 6 | 81 | 3
micrograms per liter (mcg/L)
  Cycle 2 Day 15 | -32.750 (61.6786) | -14.139 (40.4722) | 53.568 (104.0942) | 26.242 (154.4307) | 38.750 (60.3179)
  Cycle 4 Day 1: number analyzed (Participants) | 4 | 6 | 1 | 53 | 1
  Cycle 4 Day 1 | -35.500 (67.9828) | -13.967 (43.6322) | -94.000 (NA) — Standard deviation could not be estimated due to insufficient number of participants. | 3.555 (119.9087) | 10.170 (NA) — Standard deviation could not be estimated due to insufficient number of participants.
  Off-Treatment: number analyzed (Participants) | 0 | 1 | 0 | 23 | 0
  Off-Treatment |  | -3.560 (NA) — Standard deviation could not be estimated due to insufficient number of participants. |  | -22.920 (71.8744) |

20. Secondary Outcome: Phase 1 and 2: Change From Baseline in Bone Turn-over Marker - C-terminal Cross-linking Telopeptide of Type 1 Collagen (CTX)
Description: Blood samples were collected at indicated timepoint for evaluation of Bone turn-over marker CTX. Baseline is defined as the last non-missing value before the first dose of study drug (Day 1). Change from baseline was calculated as post-baseline visit value minus baseline value. Pooled data from phase 1 and phase 2 was presented for 450 mg arm as enrolled participants in both the phases had similar demographics and disease characteristics with no major changes in inclusion/exclusion criteria as defined in the protocol.
Time Frame: Baseline (predose), Cycle 2 Day 15, Cycle 4 Day 1, and off-Treatment (up to 33 months) (Cycle length = 28 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
Number analyzed (Participants) | 5 | 9 | 6 | 81 | 3
nanograms per millilitre (ng/mL)
  Cycle 2 Day 15 | 0.034 (0.1648) | 0.024 (0.1038) | -0.270 (0.3861) | 0.047 (0.4330) | -0.036 (0.1976)
  Cycle 4 Day 1: number analyzed (Participants) | 5 | 6 | 1 | 53 | 1
  Cycle 4 Day 1 | 0.028 (0.2529) | -0.008 (0.1743) | -0.549 (NA) — Standard deviation could not be estimated due to insufficient number of participants. | 0.021 (0.3562) | 0.009 (NA) — Standard deviation could not be estimated due to insufficient number of participants.
  Off-Treatment: number analyzed (Participants) | 0 | 1 | 0 | 23 | 0
  Off-Treatment |  | -0.184 (NA) — Standard deviation could not be estimated due to insufficient number of participants. |  | -0.148 (0.3735) |

ADVERSE EVENTS:
Time Frame: From start of the study up to 74 months
Description: The safety analysis set included all participants who had received at least 1 dose of study drug. As per planned analysis, pooled data for phase 1 and phase 2 for 450 mg arm was presented as enrolled participants in both the phases had similar demographics and disease characteristics. As per planned analysis the food-effect cohort of the Phase 2 only analyzed the effect of food (high-fat meal) on H3B-6545 pharmacokinetics, and no safety analyses was planned for the food-effect cohort.
Arm/Group | Phase 1: Dose Escalation: H3B-6545 100 mg | Phase 1: Dose Escalation: H3B-6545 200 mg | Phase 1: Dose Escalation: H3B-6545 300 mg | Phase 1 and Phase 2: H3B-6545 450 mg | Phase 1: Dose Escalation: H3B-6545 600 mg
All-Cause Mortality (participants affected / at risk) | 6/6 | 10/12 | 11/11 | 83/115 | 7/7
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/12 | 2/11 | 30/115 | 1/7
Other Adverse Events (participants affected / at risk) | 6/6 | 12/12 | 11/11 | 114/115 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Escalation: H3B-6545 100 mg (N=6) | Phase 1: Dose Escalation: H3B-6545 200 mg (N=12) | Phase 1: Dose Escalation: H3B-6545 300 mg (N=11) | Phase 1 and Phase 2: H3B-6545 450 mg (N=115) | Phase 1: Dose Escalation: H3B-6545 600 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alveolar lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Phase 1: Dose Escalation: H3B-6545 100 mg (N=6) | Phase 1: Dose Escalation: H3B-6545 200 mg (N=12) | Phase 1: Dose Escalation: H3B-6545 300 mg (N=11) | Phase 1 and Phase 2: H3B-6545 450 mg (N=115) | Phase 1: Dose Escalation: H3B-6545 600 mg (N=7)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (7) | 5 (5) | 39 (118) | 4 (7)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (11) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 6 (7) | 8 (8) | 52 (71) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 11 (15) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 12 (14) | 2 (2)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (4) | 3 (4) | 54 (76) | 1 (2)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (4) | 4 (4) | 4 (7) | 55 (69) | 4 (4)
Oral mucosal eruption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Tongue discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (3) | 2 (3) | 30 (48) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (4) | 4 (4) | 3 (5) | 42 (69) | 2 (6)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 2 (3) | 17 (18) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 8 (13) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thirst decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tongue fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 2 (3) | 1 (1) | 17 (25) | 0 (0)
Vestibulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginitis trichomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 1 (2) | 2 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 5 (5) | 2 (3) | 16 (32) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 5 (11) | 3 (5) | 18 (31) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 8 (9) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 10 (22) | 3 (8)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 4 (6) | 2 (2)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Blood zinc decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 13 (21) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (8) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (2) | 3 (4) | 10 (18) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroxine free increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 3 (4) | 5 (6) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 14 (15) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 2 (2) | 6 (6) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6) | 1 (2) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 1 (3)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 6 (8) | 1 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (6) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2) | 1 (1) | 2 (2) | 1 (4)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (8) | 1 (1) | 7 (10) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 3 (3) | 16 (22) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 1 (1) | 14 (16) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 8 (10) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (12) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 8 (9) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 4 (5) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (4) | 11 (21) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (7) | 1 (1) | 20 (24) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 7 (7) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 17 (18) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Neuritis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (6) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Visual perseveration (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (5) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (7) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pica (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Endometrial thickening (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Hydrometra (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2) | 1 (1) | 17 (22) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 19 (28) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (10) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 2 (2) | 3 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 17 (18) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 10 (14) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 8 (13) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Sensitive skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2/11 (2) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 3 (3) | 8 (8) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (6) | 2 (4) | 9 (14) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT03250676/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT03250676/SAP_001.pdf